CLINICAL TRIAL: NCT01912066
Title: A Phase IV Clinical Trial to Evaluate the Preventive Effectiveness of NSAID-Associated Gastroduodenal Injury (Multi-center, Double-blind, Active-controlled, Stratified Randomized, Parallel Group)
Brief Title: A Multicenter, Double Blinded, Randomized, Parallel Assignment Study to Demonstrate the Efficacy of DA9601
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DA9601_PG_IV
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: NSAID-associated Gastroduodenal Injury
MeSH Terms: interventions — DA 9601; Misoprostol; Anti-Inflammatory Agents, Non-Steroidal; aceclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stillen (Experimental): Patients taking a tab of Stillen and a tab of placebo drug and a tab of NSAID
  Interventions: Drug: Stillen; Drug: NSAID (Aceclofenac)
- Cytotec (Active Comparator): The subjects taking a tab of Cytotec, a tab of placebo drug, and a tab of NSAID
  Interventions: Drug: Cytotec (reference drug); Drug: NSAID (Aceclofenac)

INTERVENTIONS:
Drug: Stillen
  Arms: Stillen
Drug: Cytotec (reference drug)
  Arms: Cytotec
Drug: NSAID (Aceclofenac)

SUMMARY:
This is a phase IV clinical study to evaluate the preventive effectiveness of NSAID-Associated Gastroduodenal Injury. The study is consisted of multi-center, doubleblind, active-controlled, stratified randomized, parallel group. A tablet of DA9601, Cytotec (200ug of Misoprostol), Acrofen (100mg of Aceclofenac) will be assigned randomly to the subjects for four weeks.

DETAILED DESCRIPTION:
After filling an Informed consent form, subjects are joined the clinical trials. First of all, Screening test including the endoscopy test is performed.

Subjects, which fit the inclusion/Exclusion criteria, are assigned randomly. Subjects takes investigation products as randomized.

ELIGIBILITY:
Inclusion Criteria:

* Need to take NSAID pills for longer than four weeks
* should be normal diagnosed by the endoscopy test

Exclusion Criteria:

* The patients have gastric ulcer or duodenal ulcer within 30 days
* The patients have a gastro-intestinal surgery within a year
* The patients are taking the following drugs within seven days: H2 receptor antagonist, PPI, sucralfate, misoprostol, Stillen etc)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the percentage of protected subjects (%) | 4 weeks
  the definition of "protected" is the subjects with no erosions, in other words, either zero or 1 erosion found at stomach by the endoscopy.

SECONDARY OUTCOMES:
A percentage of a protected subject (at duodenum), and of ulcer occurrence | 4 weeks
  1. The definition of "protected" is the subjects with no erosions, in other words, either zero or 1 erosion found at duodenum by the endoscopy.
  2. A percentage of ulcer occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Yong Seol, MD, Study Chair — Inje University; Myoung-Gyu Choi, MD, Principal Investigator — The Catholic University of Korea; Oh Young Lee, MD, Principal Investigator — Hanyang University; Dong Ho Lee, MD, Principal Investigator — Seoul National University Bundang Hospital; Yong Chan Lee, MD, Principal Investigator — Severance Hospital; Suck Chei Choi, MD, Principal Investigator — Wonkwang University School of Medicine & Hospital; Jong Sun Rew, MD, Principal Investigator — Chonnam National University Hospital; Kang Moon Lee, Principal Investigator — Saint Vincent's Hospital, Korea; Jae Young Jang, MD, Principal Investigator — Kyunghee University Medical Center; Hoon-jai Chun, MD, Principal Investigator — Korea University Anam Hospital; Sang-woo Lee, MD, Principal Investigator — Korea University Ansan Hospital; Moo In Park, MD, Principal Investigator — Kosin University Gospel Hospital; Joong Goo Kwon, MD, Principal Investigator — Daegu Catholic University Medical Center; Geunam Song, MD, Principal Investigator — Pusan National University Hospital; Seong Woo Jeon, MD, Principal Investigator — Kyungpook National University Medical Center; Soo Taek Lee, MD, Principal Investigator — Chonbuk National University Hospital; Jae Gyu Kim, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Poong-Lyul Rhee, MD, Principal Investigator — Samsung Medical Center; Kwang Jae Lee, MD, Principal Investigator — Ajou University School of Medicine; Hyo Jin Park, MD, Principal Investigator — Gangnam Severance Hospital; Byung Ik Jang, MD, Principal Investigator — Yeungnam University Hospital; Yong Woon Shin, MD, Principal Investigator — Inha University Hospital; Dong Soo Han, MD, Principal Investigator — Hanyang University Guri Hospital; Sung Kook Kim, MD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea